CLINICAL TRIAL: NCT05300152
Title: A Comparative Evaluation of Pulpal Response to ACTIVA BioACTIVE Versus Mineral Trioxide Aggregate (MTA) As a Vital Pulpotomy Medications in Primary Teeth: an in Vivo Study
Brief Title: Pulpotomy Medications in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, shaimaa shaban mohamed el-desouky, Lecturer of Pediatric dentistry, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 398/2021
Record Dates: First submitted 2022-03-09; First posted 2022-03-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Drug Effect

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACTIVA BioACTIVE Base/Liner (Experimental): is a BioACTIVE glass-incorporated light-curable pulp capping material also known as light-cured resin-modified calcium silicate
  Interventions: Procedure: pulpotomy procedure and Histological evaluation; Diagnostic Test: Immunohistochemistry Protocol for Fibronectin Antibody; Diagnostic Test: Immunohistochemistry Protocol for Osteopontin Antibody
- Mineral trioxide aggregate (MTA) (Active Comparator): is a bioactive materials containing calcium silicate
  Interventions: Procedure: pulpotomy procedure and Histological evaluation; Diagnostic Test: Immunohistochemistry Protocol for Fibronectin Antibody; Diagnostic Test: Immunohistochemistry Protocol for Osteopontin Antibody

INTERVENTIONS:
Procedure: pulpotomy procedure and Histological evaluation — Sixty primary teeth in thirty children aged 7-9 years selected from Outpatient dental clinic Pedodontic and Endodontic Departments, Suez Canal University. divided into group I includes 30 teeth treated with ACTIVA BioACTIVE Base/Liner and group II includes 30 teeth treated by MTA with standard pulpotomy procedure Patients will be recalled after 15 and 30-days . 15 teeth from group I and 15 teeth from group II will be extracted after 15 days then subjected to decalcification then15 teeth from group I and 15 teeth from group II will be extracted after 30 days & subjected to decalcification procedure in 20% EDTA at 4 °C for approximately 5 weeks then embedded in paraffin. Serial sections will be cut at 5 µm thickness. Deparaffinize the sections by 2 changes of xylene for 10 minutes each. Stain in Harris hematoxylin solution for 8 minutes. mount with xylene based mounting medium for conventional histological assessment using light microscope
Diagnostic Test: Immunohistochemistry Protocol for Fibronectin Antibody — 1. Deparaffinization/Rehydration
     * Slides heated in an oven at 65C for 1 hour.
     * De-paraffinization
  2. Antigen Retrieval
     * Immersion of slides into staining dish containing Antigen Retrieval Solution.
     * Placing the staining dish into rice cooker.
     * When turned to warm, unplug cooker
     * Allow to cool down for 20 min
  3. Staining
     * Wash slides with TBST for 5 min on a shaker.
     * Inactivate endogenous peroxidase by 3% hydrogen peroxide for 10 min.
     * Block slides with blocking solution for 1 hour.
     * Dilute primary antibody in blocking buffer
     * Apply primary antibody to each section and incubate overnight in humidified chamber
     * Wash slides three times with TBST
Diagnostic Test: Immunohistochemistry Protocol for Osteopontin Antibody — will be carried out via avidin-biotin-peroxidase complex method using a VECTASTAIN ABC Kit . Sections will be deparaffinized by xylene and graded ethanol then treated with 20 µg/ml Proteinase K for 10 min. to prevent endogenous peroxidase activity, sections is incubated for 30 min in 0.3% H2O2/methanol then treated with 0.1% blocking serum albumin and incubated with primary antibody for 30 min. Rabbit polyclonal anti-osteopontin and goat polyclonal anti-RANKL will be used. dilution of primary antibodies used will be osteopontin (1 : 6000-8000). After being washed with phosphate-buffered saline several times, sections will be incubated with biotinylated IgG for 30 min and subsequently with streptavidin-horseradish peroxidase for 30 min. Following several washes with phosphate-buffered saline, 3,3'-diaminobenzidine substrate will be applied. As a negative control, non-immune serum will be used instead of primary antibody.

SUMMARY:
this study is aimed to evaluate and compare the pulp response to ACTIVA BioACTIVE Base/Liner and MTA as pulpotomy medication in primary teeth.

DETAILED DESCRIPTION:
Pulpotomy is an endodontic technique that involves amputating the coronal pulp and covering the residual root pulp with a clinically effective pulp medicament that is bactericidal, capable of forming a biological barrier and allows the physiological root resorption until primary tooth exfoliation. In primary dentition, pulpotomy therapy is divided into three types based on the treatment goals: devitalization (mummification), preservation, and regeneration. Formocresol is the benchmark for pulpotomy treatment in primary teeth. Buckley first used it to treat nonvital permanent teeth in 1904, and it later became a common pulpotomy medication for primary teeth primarily because of its superior clinical success and simplicity of use . However, toxicity, mutagenicity, and carcinogenicity issues posed by the possible systemic spreading of FC molecules via the root canals raised concerns on its use ; as a result, a more biocompatible, nontoxic medication was required.

Biocompatible and bioactive materials containing calcium silicate have become increasingly common in paediatric dentistry in recent years because of their properties, which include stimulation of pulp cell regeneration, re - routing of the inflammatory response, and improving the healing ability of the remaining vital pulp . Mineral trioxide aggregate (MTA) was developed and implemented as a root-end filling at Loma Linda University in California, USA, in 1993; its physical and chemical properties were identified by Torabinejad et al ., in 1995. MTA is a chemical compound composed of tricalcium silicate, dicalcium silicate, tricalcium aluminate, calcium sulphate dehydrate, gypsum, and bismuth oxide . It hydrates to form a colloidal gel with a pH of 12.5, equivalent to that of calcium hydroxide . Moreover, it takes 3 to 4 hours to set with a compressive strength of 70 Mpa after setting, which is comparable to Intermediate Restorative Material (IRM) . MTA is a biocompatible substance that seals better than amalgam or zinc oxide eugenol (ZOE) [30-32] also, it retains pulp vitality and induces repair as it comes into contact with dental pulp or peri-radicular tissues. MTA has been thoroughly examined clinically and radiologically, as well as compared to other pulpotomy medicaments, and it has been reported that MTA should be considered the new gold standard for pulp-capping therapy. On the other hand, MTA has some drawbacks, including difficulty in manipulation, a long setting duration, a high cost, poor mechanical properties, poor adhesion to dental tissue and tooth staining .

Several recent calcium silicate-based materials have been developed in order to alleviate MTA's drawbacks. ACTIVA BioACTIVE Base/Liner, a BioACTIVE glass-incorporated light-curable pulp capping material, was recently introduced in 2014 as a "light-cured resin-modified calcium silicate" (RMCS) claiming composite's resilience, aesthetics, and physical properties, as well as improved calcium, phosphate, and fluoride release when compared to glass ionomer . It comprised of a diurethane and methacrylate-based monomer with a modified polyacrylic acid and polybutadiene-modified diurethane dimethacrylate as well as BioACTIVE glass as a filler . ACTIVA has three setting reactions: it cures with low intensity light for 20 seconds per layer and has both glass-ionomer (acid-base reaction) and composite self-cure setting reactions. The bioactivity of ACTIVA BioACTIVE products is dependent on a process in which the material reacts to pH cycles and actively participates in the release and recharging of considerable amounts of calcium, phosphate, and fluoride . Theses mineral components are concerned with promoting the development of mineralized hard tissue also, they promote the creation of a connective apatite layer and the development of a seal at the material-tooth interface .

ELIGIBILITY:
Inclusion Criteria:

* Healthy & cooperative child
* No history of spontaneous pain
* No pathologic tooth mobility
* Normal gingival and periodontal condition
* Absence of furcal/periapical radiolucency

Exclusion Criteria:

* Uncooperativeness of child and/or parents
* Unrestorable tooth
* history of spontaneous pain
* Percussion sensitivity

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
the regenerative effect of ACTIVA BioACTIVE Base/Liner and MTA as pulpotomy medication in primary teeth | 12 months
  by assessment of reparative dentin formation in the histological sections of the tested teeth by detection of the presence of odontoblast cells (dentin forming- cells) and mineralized tissue between the capping material and the remaining pulp tissue.

SECONDARY OUTCOMES:
the reparative dentinogenesis process after application of ACTIVA BioACTIVE Base/Liner and MTA as pulpotomy medication in primary teeth | 12 months
  by assessment the molecular signalling (production of fibronectin & osteopontin antibody) involved in cell differentiation during reparative dentinogenesis process using Immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
protocol & conclusion
Supporting Information: Study Protocol, SAP
Time Frame: for 1 month
URL: http://suez.edu.eg

REFERENCES:
- [Background] Holan G, Eidelman E, Fuks AB. Long-term evaluation of pulpotomy in primary molars using mineral trioxide aggregate or formocresol. Pediatr Dent. 2005 Mar-Apr;27(2):129-36. PMID 15926290
- [Background] Gandolfi MG, Siboni F, Prati C. Chemical-physical properties of TheraCal, a novel light-curable MTA-like material for pulp capping. Int Endod J. 2012 Jun;45(6):571-9. doi: 10.1111/j.1365-2591.2012.02013.x. Epub 2012 Mar 31. PMID 22469093
- [Background] Anthoney D, Zahid S, Khalid H, Khurshid Z, Shah AT, Chaudhry AA, Khan AS. Effectiveness of Thymoquinone and Fluoridated Bioactive Glass/Nano-Oxide Contained Dentifrices on Abrasion and Dentine Tubules Occlusion: An Ex Vivo Study. Eur J Dent. 2020 Feb;14(1):45-54. doi: 10.1055/s-0040-1703418. Epub 2020 Mar 13. PMID 32168531
- [Background] Avram DC, Pulver F. Pulpotomy medicaments for vital primary teeth. Surveys to determine use and attitudes in pediatric dental practice and in dental schools throughout the world. ASDC J Dent Child. 1989 Nov-Dec;56(6):426-34. PMID 2530256
- [Derived] Omer SMM, Elsaied HAF, Alghonemy WY, El-Desouky SS. Histopathological and immunohistochemical characterization of pulp tissue reaction to ACTIVA BioACTIVE base/liner in primary teeth pulpotomy: a randomized clinical trial. BMC Oral Health. 2025 Jun 3;25(1):885. doi: 10.1186/s12903-025-06177-x. PMID 40457274